CLINICAL TRIAL: NCT01264237
Title: An Enriched Enrollment, Double-Blind, Placebo-Controlled, Parallel Group, Randomized Withdrawal Trial to Evaluate the Efficacy, Tolerability and Safety of Etoricoxib (Arcoxia) in Patients With Moderate to Severe Neuropathic Pain
Brief Title: Evaluation of the Efficacy, Tolerability and Safety of Etoricoxib (Arcoxia) in Patients With Neuropathic Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Analgesic Solutions (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Stuart Ratcliffe, MBChB, MFPM, FRSM. Director of Pain Research, MAC UK Neuroscience Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRK008b-2010
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Postherpetic Neuralgia; Neuralgia
Keywords: Postherpetic neuralgia; Neuropathic pain; Etoricoxib
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etoricoxib (Experimental): The study will use an Enriched Enrollment Randomized Withdrawal (EERW) design consisting of a 2-week open-label enrichment phase, during which subjects will receive etoricoxib. Patients who experience at least a 30% reduction in pain intensity will be randomized to either continued treatment with etoricoxib 90 mg qd or matching placebo (at a 1:1 ratio) for 4 weeks.
  Interventions: Drug: Etoricoxib
- Placebo (Placebo Comparator): The study will use an Enriched Enrollment Randomized Withdrawal (EERW) design consisting of a 2-week open-label enrichment phase, during which subjects will receive etoricoxib, followed by a 4-week randomized, double-blind, placebo-controlled treatment phase, during which subjects will receive either etoricoxib or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etoricoxib — 90mg Tablet QD at 10:00a.m.
  Other Names: Arcoxia
  Arms: Etoricoxib
Drug: Placebo — One tablet QD at 10:00a.m.
  Arms: Placebo

SUMMARY:
The present study will aim to determine the safety, efficacy, and tolerability of etoricoxib, an NSAID pain reliever, in patients with Neuropathic pain. Neuropathic pain, or pain caused by abnormal activity of sensory neurons, remains undertreated. Post herpetic neuralgia (PHN), which is commonly referred to as post-shingles pain, is the most useful disease to study when investigating the efficacy of pain relievers for Neuropathic pain. Therefore, this study will primarily involve patients with PHN.

The hypothesis in this study is that etoricoxib efficacy is superior to that of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Be a man or a non-pregnant, non-lactating woman 18 years and older. Women of childbearing potential should be willing to use an acceptable birth control method (at the investigator's discretion) during the study to avoid pregnancy.
* Have voluntarily provided written informed consent.
* Be able to speak, read, write, and understand English, understand the consent form, complete study related procedures, and communicate with the study staff.
* Have a clinical diagnosis of PHN by history or objective findings in the opinion of the Investigator for a minimum of 6 months. If the patient pool needs to be expanded to other neuropathic conditions, patients must meet the same criteria of patients with PHN and in addition must have a clinical diagnosis of peripheral diabetic neuropathy (PDN), idiopathic sensory neuropathy (ISN) or small fiber predominant neuropathy (SFN) by history or clinical findings in the opinion of the investigator for a minimum of 6 months.
* Have a pain intensity score averaging ≥3 on a 0-10 NRS for average daily recall over past 24 hours (at Visit 1)
* Be, in the opinion of the investigator, in generally good health (other than PHN) at screening, based upon the results of a medical history, physical examination and laboratory analysis

Exclusion Criteria:

* Are pregnant and/or lactating
* Have been diagnosed as having any inflammatory arthritis, gout, pseudo-gout, Paget's disease, fibromyalgia or any chronic pain syndrome that in the Investigator's opinion would interfere with the assessment of pain and other symptoms of PHN
* Have evidence for multiple causes of pain in the neuropathic pain area, such as lumbar radiculopathy in an area of lumbosacral PHN
* Have any bodily moderate to severe pain (e.g., osteoarthritis) that could confound assessment or self-evaluation of pain due to PHN
* Use NSAID compounds (oral and topical) within 1 week of study and for the duration of the study
* Use opioids including tramadol within 1 week of study and for the duration of the study. (Other NP medications are allowed, provided that the doses have been stable for at least one month prior to Visit 1)
* Have had neuro-ablation or neurosurgical intervention for their PHN
* Have received nerve block or intrathecal analgesia within 6 weeks of study
* Have a history of congestive heart failure, unstable coronary artery disease, stroke, or uncontrolled hypertension
* Have a history of significant gastrointestinal disease, including active gastro-duodenal ulcerations, perforations, or bleeds
* Have abnormal clinical laboratory test results or vital signs unless deemed not clinically significant by the investigator
* Have skin lesions or damage in the area where BSTK measurements are conducted (only applicable to PHN patients)
* Are undergoing active treatment for cancer, are known to be infected by HIV, or are being acutely and intensively immunosuppressed following transplantation
* Have a history of alcohol or other substance abuse (not including nicotine or tobacco) within five years
* Known to have a condition that in the investigator's judgment precludes participation in the study
* Have a significant psychiatric disorder in the opinion of the Investigator.
* Have received an investigational drug or have used an investigational device in the 30 days prior to study entry
* Have previously been admitted to this study
* Are allergic to Arcoxia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-08 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Time to Efficacy Failure | 28 Days
  To compare the efficacy of etoricoxib to placebo in reducing pain intensity in patients with NP, as measured by Time to Efficacy Failure during the Double-Blind Period.

SECONDARY OUTCOMES:
To evaluate the efficacy of etoricoxib in NP during the Open-Label and the Double-Blind Periods | 42 Days
Time to efficacy failure by PHN sub-group based on sensory testing results | 42 Days
Safety as assessed by adverse events, serious adverse events, and vital signs | 56 Days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Ratcliffe, MBChB, MFPM, FRSM, Principal Investigator — MAC (UK) Neuroscience Ltd
Locations (2):
- United Kingdom (2):
  - MAC (UK) Neruoscience Ltd, Liverpool
  - MAC (UK) Neuroscience Ltd, Manchester